CLINICAL TRIAL: NCT04648098
Title: The Effect of Post-stroke Discharge Training and Telephone Counseling Service on Patients' Functional Status and Caregiver Burden: A Randomised Control Trial
Brief Title: Effect of Post-stroke Discharge Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Collaborators: Trakya University (Other)
Responsible Party: Principal Investigator, Deniz Ezgi Bitek, Principal Investigator, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: interventional
Record Dates: First submitted 2020-11-18; First posted 2020-12-01 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Caregiver Burnout
MeSH Terms: conditions — Stroke; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention group (Experimental): Discharge training and telephone counseling
  Interventions: Other: Discharge training and telephone counseling
- No Intervention: Control Group (No Intervention): Routine care

INTERVENTIONS:
Other: Discharge training and telephone counseling — The discharge training was given by using different teaching methods in the form of verbal expression, demonstration, and question and answer. The care guide prepared by the researchers in line with the literature was used as a training material for stroke patients and their caregivers.The training varied according to the learning level of individuals but took an average of 40-60 minutes.
  Consultation service was given to the caregivers one week after discharge and once a month for three months by telephone call.
  Arms: Experimental: Intervention group

SUMMARY:
The aim of this study was to determine the effect of post-stroke discharge training and telephone counseling service on patients' functional status and caregiver burden. The study was conducted with 69 stroke patients (34 in the intervention group and 35 in the control group) and their caregivers. In the study, data were collected before discharge and three months after discharge. Discharge training and telephone counseling (one week after discharge and once a month for three months) were given to the caregivers of the patients in the intervention group.

DETAILED DESCRIPTION:
This study, which was planned as a randomised controlled study, was conducted university hospital neurology clinic in Turkey. A total of 80 participants who met the inclusion criteria were randomised to either the intervention and control groups.

In this study, Patient Information Form, Modified Rankin Scale and Barthel Index were used to collect data about patients, while Caregiver Information Form and Caregiver Burden Scale were used to collect data about caregivers Pre-tests were applied to patients and caregivers in the intervention and control groups before discharge. After the pre-tests were applied to the caregivers in the intervention group, discharge training was given.

ELIGIBILITY:
Inclusion Criteria:

* the age of 18 and over (for patients and caregivers)
* having undergone a hemorrhagic or ischemic stroke (for patients)
* being literate (for caregivers)
* being primarily responsible for the care of the stroke patient during the hospital stay and at home after discharge (for caregivers)
* using a mobile or home phone (for caregivers)
* being open to communication and collaboration (for caregivers)

Exclusion Criteria:

* Rankin Scale score of 4 above (for patients)
* Having problem in terms of hearing and understanding (for caregivers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Caregiver Burden Scale | Change from baseline score at the end of the third month
  Caregiver Burden Scale, developed by Zarit et al. (1980), was used to evaluate the care burden of patient relatives. There are 22 expressions in the scale that determine the effect of caregiving on the individual's life. The score obtained from the five-point Likert scale is minimum 0 and maximum 88.A high score on the scale indicates that the problem experienced by the caregiver is high.
The Barthel Index | Change from baseline score at the end of the third month
  The Barthel Index to developed by Mahoney and Barthel in 1965 to evaluate physical independence in daily life activities. Index consists of 10 items that include daily life activities and is used to evaluate the level of functional independence. Items in the scale are graded between 0 and 15 points in 5 increments according to the question. The score ranges from 0 to 100 (0-20 points fully dependent, 21-61 points highly dependent, 62-90 points moderately dependent, 91-99 points slightly dependent, 100 points fully independent).
Modified Rankin Scale | Change from baseline score at the end of the third month
  Modified Rankin Scale evaluating the functional limitation and degree of addiction occurring in the patient after stroke was evaluated in seven categories (0: No symptoms, 1: No obvious deficits, 2: Mild deficits, 3: Moderate deficits, 4: Severe deficits, 5: Very severe deficit and 6: Death).

CONTACTS AND LOCATIONS:
Overall Officials: Özgül EROL, Study Director — Trakya University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No